CLINICAL TRIAL: NCT03834324
Title: The Effects of FES Cycling Combined With Virtual Reality Racing on Lower Limb Voluntary Function After Incomplete SCI: A Pilot Study.
Brief Title: Functional Electrical Stimulation During Cycling in People With Spinal Cord Injury
Acronym: iCycle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: University College, London (Other)
Responsible Party: Principal Investigator, Jane Burridge, PhD, Professor of Restorative Neuroscience, University of Southampton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6054
Record Dates: First submitted 2019-02-05; First posted 2019-02-07 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2019-02

CONDITIONS: Spinal Cord Injuries
Keywords: Functional Electrical Stimulation; Cycling; Virtual Reality
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Technology development and Observational study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention (Experimental): FES
  Interventions: Device: FES

INTERVENTIONS:
Device: FES — Functional Electrical Stimulation during cycling with Virtual Reality Feedback

SUMMARY:
Neuroscience research that has identified potential for recovery (neuroplasticity) following incomplete SCI has changed clinical practice away from compensation strategies towards optimizing recovery. Important factors include: repetitive exercise, Functional Electrical Stimulation (FES) and appropriate feedback. The iCycle combines repetitive exercise with FES and provides feedback on performance in a virtual cycle race. Unlike previous devices, performance in the race is determined only by voluntary effort (i.e. not torque generated by FES plus voluntary effort). In this study with incomplete SCI participants we will test the iCycle with six inpatients to refine the protocol and make technical improvements. We will then conduct an ABA pilot study (n=10) in which a 3G-connected iCycle is used in people's own homes. We will compare usual care (A) with iCycle exercise (B). Changes in neural connectivity (TMS evoked EMG potentials), muscle strength and walking will be measured as well qualitative analysis of users' views.

DETAILED DESCRIPTION:
Background: Functional Electrical Stimulation (FES) cycling can benefit health and may lead to neuroplastic changes following incomplete spinal cord injury (SCI). Our hypothesis is that greater neuroplastic effects occur when electrical stimulation of peripheral nerves is combined with voluntary drive. In this pilot study, we will investigate the effects of a one-month training programme using a novel device, the iCycle, in which voluntary effort (cortical drive) is encouraged by virtual reality biofeedback during FES cycling.

Methods: Eleven participants (C1-T12) with incomplete SCI (5 sub-acute; 6 chronic) will be recruited and undergo 12-sessions of iCycle training. Function will be assessed before and after training using the bilateral ISNC-SCI motor score neurological (motor) function, Oxford power grading, Modified Ashworth Score, Spinal Cord Independence Measure, the Walking Index for Spinal Cord Injury and 10m-walk test. Power output will be measured during training.

ELIGIBILITY:
Inclusion Criteria:

1. using a wheelchair for at least two hours per day

Exclusion Criteria:

1. cardiac pacemaker
2. pressure sores or unresolved skin problems
3. unhealed lower limb fractures
4. pregnancy
5. active heterotrophic ossification (lower limbs)
6. severe osteoporosis
7. complex regional pain syndrome
8. metal implants near electrode sites
9. lower limb malignancy
10. T6 and below spinal malignancy
11. uncontrolled autonomic dysreflexia
12. history of knee dislocation/subluxation
13. allergy to electrodes
14. cognitive difficulties
15. severe spasticity (Ashworth scale 4 or 5 in muscle groups that would prevent smooth pedalling) or
16. neurological degenerative diseases.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-05-03 (Actual); Primary Completion 2016-04-29 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
International Standards for Neurological Classification of Spinal Cord Injury (ISNC-SCI). | Change between baseline and 4 weeks
  Neurological Classification
International Standards for Neurological Classification of Spinal Cord Injury (ISNC-SCI). | Change between baseline and 8 weeks
  Neurological Classification

SECONDARY OUTCOMES:
Oxford scale motor power grading | Change between baseline and 4 weeks
  Muscle strength
Oxford scale motor power grading | Change between baseline and 8 weeks
  Muscle strength
Modified Ashworth Score (MAS) | Change between baseline and 4 weeks
  Spasticity / stiffness
Modified Ashworth Score (MAS) | Change between baseline and 8 weeks
  Spasticity / stiffness
Spinal Cord Independence Measure (SCIM) | Change between baseline and 4 weeks
  ADL
Spinal Cord Independence Measure (SCIM) | Change between baseline and 8 weeks
  ADL
Walking Index for Spinal Cord Injury (WISCI II) | Change between baseline and 4 weeks
  Walking ability
Walking Index for Spinal Cord Injury (WISCI II) | Change between baseline and 8 weeks
  Walking ability

CONTACTS AND LOCATIONS:
Overall Officials: Trudi Bartlett, BSc, Study Chair — University of Southampton

IPD SHARING:
Plan to Share IPD: No
we have no specific plan for this

REFERENCES:
- [Result] Duffell LD, Paddison S, Alahmary AF, Donaldson N, Burridge J. The effects of FES cycling combined with virtual reality racing biofeedback on voluntary function after incomplete SCI: a pilot study. J Neuroeng Rehabil. 2019 Nov 27;16(1):149. doi: 10.1186/s12984-019-0619-4. PMID 31771600